CLINICAL TRIAL: NCT04837131
Title: A Phase 2 Open-Label Pilot Study of the Safety and Tolerability of Ixazomib Administered Orally to Patients With Scleroderma-Related Interstitial Lung Disease
Brief Title: A Study to Evaluate the Safety and Tolerability of Oral Ixazomib in Scleroderma-related Lung Disease Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Michael M. Pham (Other)
Responsible Party: Sponsor-Investigator, Michael M. Pham, Regulatory Sponsor and Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-004201
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Systemic Sclerosis; Scleroderma; Diffuse Systemic Sclerosis; Diffuse Scleroderma; Diffuse Cutaneous Systemic Sclerosis; Diffuse Cutaneous Scleroderma; Progressive Systemic Sclerosis; Progressive Scleroderma; Scleroderma, Systemic; Scleroderma, Diffuse; Scleroderma;Progressive; Systemic Sclerosis, Diffuse; Systemic; Sclerosis, Progressive; Scleroderma of Lung; Scleroderma With Pulmonary Involvement; Systemic Sclerosis Pulmonary; Systemic Sclerosis With Lung Involvement; Interstitial Lung Disease; Pulmonary Fibrosis Interstitial
Keywords: Scleroderma; Systemic Sclerosis; Interstitial Lung Disease; Ixazomib; Mycophenolate; Treatment
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Lung Diseases, Interstitial; Pulmonary Fibrosis | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ixazomib in patients with scleroderma-interstitial lung disease (ILD) (Experimental): Participants will be administered oral ixazomib for six cycles (each cycle is 28 days duration).
  Interventions: Drug: Ixazomib

INTERVENTIONS:
Drug: Ixazomib — Ixazomib 4 mg capsule taken orally on days 1, 8, and 15 of a 28-day treatment cycle repeated for 6 cycles

SUMMARY:
The purpose of this research study is to learn about the effects of the medication ixazomib in participants with scleroderma/systemic sclerosis including its safety and tolerability, its effects on skin, lungs and other organs, and its effects on overall health and quality of life.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety and tolerability of oral ixazomib taken on days 1, 8, and 15 of each 28-day treatment cycle for 6 cycles in 12 participants having diffuse systemic sclerosis/scleroderma of less than 5 years duration with non-severe interstitial lung involvement as identified from chest CT scan completed within the preceding 3 months or at study screening visit. All 12 participants will receive oral ixazomib. Reflecting the common use of mycophenolate in the management of scleroderma with complicating interstitial lung disease, 6 of 12 participants who will be enrolled will be already taking mycophenolate at a stable dose for the preceding 3 months and will be allowed to continue taking mycophenolate throughout the entire study prescribed as routine care. Ixazomib will be added to their medications. The remaining 6 of 12 participants meeting the same eligibility criteria will not be using mycophenolate or any other treatment for scleroderma interstitial lung disease at the time of enrollment and will subsequently take ixazomib study medication during participation in this study. Ixazomib dose modification or interruption is allowed for safety and tolerability reasons at any time during the study.

The secondary objective of this study is to assess the effect of ixazomib on scleroderma skin tightness/thickening and its effect on scleroderma interstitial lung disease.

The study includes approximately 13 clinic visits over up to approximately 10 months. Study procedures include medical examinations, blood tests, chest CT scans, pulmonary function tests, echocardiogram, EKG, skin biopsies, and questionnaires.

There is no cost for participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, age ≥18 years at time of signing informed written consent
* Confirmed diagnosis of diffuse cutaneous systemic sclerosis/scleroderma
* Disease duration not longer than 60 months defined as the time from the first non-Raynaud phenomenon manifestation
* Scleroderma skin thickness score (modified Rodnan skin score) between 15 and 45
* Evidence of scleroderma-related lung involvement on chest CT scan completed within the preceding 3 months or at screening study visit
* Pulmonary function testing demonstrating FVC ≥45% predicted and DLCO ≥40% predicted at screening study visit
* Resting transthoracic echocardiogram within the preceding 6 months or at screening study visit without evidence of pulmonary artery hypertension
* Stable mycophenolate dose during the preceding 3 months for those who are taking mycophenolate. Mycophenolate use is not an eligibility requirement to participate; but those participants already using mycophenolate at screening study visit will continue taking the medication throughout the entire study.
* Willingness to undergo supervised withdrawal during the first 90 days of the study of any other medication besides mycophenolate used specifically as treatment of scleroderma-related interstitial lung disease with confirmed stable pulmonary status.
* Willingness to undergo supervised withdrawal during the first 90 days of the study of any other prohibited medications with confirmed stable status.
* Able to understand and sign a written informed consent form
* Able to understand the importance of adhering to study treatment and the study protocol, and willing and able to follow all study requirements, including the concomitant medication restrictions, throughout the study
* Practice birth control requirements for sexually active female participants including option of abstinence for the entire study and for at least 90 days after the last dose of study medication
* Practice birth control requirements for sexually active male participants or partners including option of abstinence for the entire study and for at least 90 days after the last dose of study medication

Exclusion Criteria:

* Pulmonary artery hypertension under treatment
* Evidence of clinically significant pulmonary hypertension or left ventricular dysfunction with left ventricular ejection fraction < 40% from either prior heart catheterization or resting transthoracic echocardiography within the preceding 6 months.
* Evidence of significant gastrointestinal involvement by scleroderma as assessed by the University of California, Los Angeles, Scleroderma Clinical Trial Consortium Gastrointestinal Tract multi-item questionnaire, 2.0 ([UCLA SCTC GIT 2.0) at screening study visit.
* Known esophageal stricture sufficient to limit the ability to swallow oral medication
* Prior history of scleroderma renal crisis
* Another connective-tissue disorder (eg, rheumatoid arthritis, systemic lupus erythematosus)
* Any other significant pulmonary disorder (e.g., chronic obstructive pulmonary disease, emphysema, adult moderate to severe asthma)
* Significant environmental exposure known to cause pulmonary fibrosis including, but not limited to, drugs (e.g., amiodarone), asbestos, beryllium, radiation, or domestic birds or other exposures associated with hypersensitivity pneumonitis
* Unstable or deteriorating cardiac disease within the preceding 6 months including but not limited to unstable angina pectoris, myocardial infarction (heart attack), heart failure requiring hospitalization, poorly controlled heart arrhythmia, or significant pericardial effusion/fluid collection around the heart
* Known liver disease (e.g., chronic hepatitis or cirrhosis)
* Significant abnormality of liver function tests
* Significant kidney function impairment of any cause as evidenced by creatinine clearance <30 mL/min
* Known active or suspected peptic (stomach) ulcer
* Known active hematologic blood-related disorder other than anemia of chronic disease or iron deficiency anemia
* Significant abnormality of blood count including hemoglobin ≤ 8.0 gm/dl, absolute neutrophil count ≤ 1000, or platelet count ≤ 75,000
* Known hematologic blood-related malignancy
* Prior stem cell or bone marrow transplant
* History of any malignancy within the last 5 years other than non-melanoma skin cell cancer cured by local resection or a carcinoma-in-situ
* Any condition likely to result in death within 12 months.
* Any condition which might be significantly worsened by the known side effects associated with ixazomib including known ≥ grade 2 peripheral neuropathy
* Tobacco smoking within 3 months of screening study visit or unwillingness to avoid smoking throughout the study (e.g., cigarette, pipe, or cigar)
* History of alcohol or substance abuse in the previous 2 years
* Any active infection including, but not limited to, bronchitis, pneumonia, sinusitis, or urinary tract infection
* Pregnancy or lactation/breast feeding
* Expectation of study participation being interrupted on account of a foreseeable medical or surgical event
* Prior use of ixazomib or other proteasome inhibitor medication
* Suspected intolerance, allergy, or hypersensitivity to ixazomib or any of its excipients
* Any prior use of rituximab
* Any prior use of cyclophosphamide
* Ongoing use within the preceding 28 days or expected use of an investigational drug (an investigational drug is defined as any drug that has not been FDA approved for marketing)
* Ongoing use or expected use of any of the following therapies: Strong inducers of a cytochrome drug metabolizing enzyme in the liver (CYP3A ). (e.g. rifampin, rifapentine, rifabutin, carbamazepine, enzalutamide, phenytoin, fosphenytoin, phenobarbital, St. John's wort)
* Ongoing use or expected use of any of the following medications: cyclophosphamide, rituximab, abatacept, nintedanib, tocilizumab, intravenous immunoglobulin (IVIG), methotrexate, leflunomide, azathioprine, sirolimus, tacrolimus, oral corticosteroids at a dose >10 mg/d prednisone equivalent, D-penicillamine, minocycline, interferon-γ, bosentan, ambrisentan, macitentan, phosphodiesterase inhibitors (sildenafil or tadalafil for uses other than erectile dysfunction or Raynaud phenomenon), riociguat, tumor necrosis factor-α (TNF-α) inhibitors (infliximab, etanercept, adalimumab, certolizumab, golimumab), and cyclosporine, .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pham, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study to Evaluate the Safety and Tolerability of Oral Ixazomib in Scleroderma-related Lung Disease Patients — https://www.mayo.edu/research/clinical-trials/cls-20508101

RESULTS

PARTICIPANT FLOW:
Groups:
- Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD): Participants were administered oral ixazomib for six cycles (each cycle is 28 days duration).
  Ixazomib: Ixazomib 4 mg capsule taken orally on days 1, 8, and 15 of a 28-day treatment cycle repeated for 6 cycles
Period: Overall Study
Arm/Group | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD)
Started | 4
Completed | 0
Not Completed | 4
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD)
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (23.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Event (AE)
Description: The number of participants with at least one treatment-emergent adverse event. Defined as any of the following: Treatment-emergent AEs; Treatment-emergent serious adverse events (SAEs); Treatment-emergent treatment-related AEs; or Treatment-emergent treatment-related SAEs.
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD)
Number analyzed (Participants) | 3
Participants | 3

2. Primary Outcome: Adverse Events Leading to Ixazomib Dose Modifications
Description: Number of participants with treatment-emergent AEs leading to ixazomib dose modifications.
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD)
Number analyzed (Participants) | 3
Participants | 2

3. Primary Outcome: Adverse Events Leading to Ixazomib Early Discontinuation
Description: Number of participants with treatment-emergent AEs leading to ixazomib early discontinuation.
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD)
Number analyzed (Participants) | 3
Participants | 2

4. Primary Outcome: Change in the UCLA Scleroderma Clinical Trials Consortium Gastrointestinal 2.0 (UCLA SCTC GIT 2.0) Questionnaire Score
Description: The UCLA SCTC GIT 2.0 is a self-administered survey consisting of 34 questions (Reflux 1 to 8, Distention/Bloating 9 to 12, Fecal Soilage 13, Diarrhea 14 to 15, Social functioning 16 to 21, Emotional well-being 22 to 30, Constipation 31 to 34). The items are scored on a scale from 0 to 3, where 0 indicates better health and 3 indicates worse health, except for questions 15 and 31, which are scored as 0 (better health) and 1 (worse health). Scores from all scales except the constipation scale are averaged to form a total GIT score from 0 (no gastrointestinal problems) to 3 (most severe) that captures overall burden of severity of scleroderma-associated gastrointestinal involvement.
Time Frame: Baseline, 7 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD)
Number analyzed (Participants) | 3
score on a scale | -0.09 (0.156)

5. Secondary Outcome: Change From Baseline in Modified Rodnan Skin Score (MRSS)
Description: MRSS is a validated clinical semiquantitative assessment of scleroderma skin thickness at 17 prespecified sites on the body, with thickness at each site scored from 0 (uninvolved) to 3 (severe thickening) that are tabulated for a total numerical skin score ranging 0-51. Lower scores indicate less involvement, and higher scores indicate more severe thickening.
Time Frame: Baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD)
Number analyzed (Participants) | 3
score on a scale | -4.33 (11.02)

6. Secondary Outcome: Change From Baseline in High Resolution Chest CT Scan Goh Score
Description: Staging extent of scleroderma lung involvement on high resolution chest CT scan by the application of Goh criteria which identified a severity extent threshold of 20% lung involvement yields two cohorts with significantly different 10 year survivorship. Goh scores range 0-100% with a higher score indicating greater extent of lung involvement.
Time Frame: Baseline, 24 weeks
Population: Chest CT scan not performed on any participants. Data not collected nor analyzed as study was terminated due to low enrollment.
Arm/Group | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD)
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in Forced Vital Capacity (FVC) % Predicted.
Description: FVC is the maximum amount of air a person can forcefully exhale from their lungs after taking a deep breath.
Time Frame: Baseline, 7 months
Measure: Mean (Standard Deviation); unit: percentage of air
Arm/Group | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD)
Number analyzed (Participants) | 3
percentage of air | -0.33 (5.51)

8. Secondary Outcome: Change in Total Lung Capacity (TLC) % Predicted
Description: TLC is the total maximum amount of air that lungs can hold.
Time Frame: Baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: percentage of air in lungs
Arm/Group | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD)
Number analyzed (Participants) | 2
percentage of air in lungs | 5 (39.11)

9. Secondary Outcome: Severity of Dyspnea at Baseline (Mahler Baseline Dyspnea Index)
Description: Severity of dyspnea at baseline is measured with the Mahler Baseline Dyspnea Index (BDI). BDI includes 5 grades of severity from 0 (severe impairment) to 4 (no impairment ) for each of 3 categories (functional impairment; magnitude of task; magnitude of effort) yielding a summation focal score (0-12). Higher scores indicate lower impairment.
Time Frame: Baseline
Population: Mahler Baseline Dyspnea Index was not completed by any subject. Data not collected nor analyzed as study was terminated due to low enrollment.
Arm/Group | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD)
Number analyzed (Participants) | 0

10. Secondary Outcome: Dyspnea Status Rating (Mahler Transitional Dyspnea Index)
Description: Mahler Transitional Dyspnea Index (TDI) rates a participant's dyspnea status relative to baseline. TDI scores range from -3 (major deterioration) to +3 (major improvement) including 0 to indicate no change in status for each of the 3 BDI categories (functional impairment; magnitude of task; magnitude of effort) yielding a summation focal score (-9 to +9). Higher scores indicate major improvement.
Time Frame: 12 weeks, 24 weeks
Population: Mahler Transitional Dyspnea Index was not completed by any subject. Data not collected nor analyzed as study was terminated due to low enrollment.
Arm/Group | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD)
Number analyzed (Participants) | 0

11. Secondary Outcome: Change in Scleroderma Health Assessment Questionnaire (SHAQ) Score
Description: SHAQ self-assesses function in 8 domains of the Health Assessment Questionnaire Disability Index (HAQ-DI): dressing and grooming, arising, eating, walking, hygiene, reach, grip, and activities. Highest domain scores 0 (no difficulty) to 3 (unable to do) are summed and divided by 8 to yield Disability Index score as a continuous variable ranging 0 to 3.
  SHAQ has:1) a 15-cm Visual Analog Scale (VAS) rating pain with anchors "No Pain" and "Very Severe Pain"; 2) four 15-cm VAS assessing Raynaud phenomenon, digital ulcers, gastrointestinal and lung symptoms with anchors "Does Not Interfere" and "Very Severe Limitation"; and 3) overall disease severity 15-cm VAS with anchors "No Disease" and "Very Severe Disease"
Time Frame: Baseline, 24 weeks
Population: Scleroderma Health Assessment Questionnaire was not completed by any subject. Data not collected nor analyzed as study was terminated due to low enrollment.
Arm/Group | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD)
Number analyzed (Participants) | 0

12. Secondary Outcome: Change in Patient Global Assessment of Disease Activity (PtGA)
Description: Patient-reported outcome that represents the participant's assessment of his or her current overall health (Question: How was your overall health in the last week?) rated on an 11-point numeric scale anchored at 0 (excellent) to 10 (extremely poor) with higher scores indicating worse disease in terms of severity and damage.
Time Frame: Baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD)
Number analyzed (Participants) | 2
score on a scale | 3.4 (3.3)

13. Secondary Outcome: Change in Physician Global Assessment of Disease Activity (MDGA)
Description: Physician-reported outcome that represents an assessment of the participant's current overall health rated on an 11-point numeric scale anchored at 0 (excellent) to 10 (extremely poor) with higher scores indicating worse disease in terms of severity and damage.
Time Frame: Baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD)
Number analyzed (Participants) | 3
score on a scale | 1.7 (1.0)

14. Secondary Outcome: Change in American College of Rheumatology Composite Response Index for Clinical Trials in Early Diffuse Cutaneous Systemic Sclerosis (ACR CRISS)
Description: ACR CRISS calculates the predicted probability of improvement in a 2-step process.
  Four possible outcomes in Step 1 include worsening of FVC % predicted by at least 15%, new decline of left ventricular ejection fraction to 45% or less attributable to scleroderma and needing treatment, new onset pulmonary arterial hypertension attributable to scleroderma and scleroderma renal crisis. If any one of these outcomes develops as a change from baseline, the participant is classified as not improved (score = 0) regardless of changes in other parameters.
  Step 2 calculates change from baseline in the predicted probability of improvement based on combined changes in the mRSS, FVC % predicted, patient global assessment, physician global assessment, and HAQ-DI. The calculated probability ranges from 0 (not improved) to 1.0 where a higher score indicates improvement.
Time Frame: Baseline, 24 weeks
Population: American College of Rheumatology Composite Response Index testing was not completed by any subject. Data not collected nor analyzed as study was terminated due to low enrollment.
Arm/Group | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD)
Number analyzed (Participants) | 0

15. Secondary Outcome: Change in Diffusion Capacity (DLCO) % Predicated
Description: DLCO is the amount of carbon monoxide (CO) that moves from the lungs to the blood
Time Frame: Baseline, 7 months
Measure: Mean (Standard Deviation); unit: percentage of carbon monoxide
Arm/Group | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD)
Number analyzed (Participants) | 3
percentage of carbon monoxide | 0 (5.30)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to completion of the post-treatment follow-up visit, approximately 16 months.
Arm/Group | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD)
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixazomib in Patients With Scleroderma-interstitial Lung Disease (ILD) (N=4)
Pruritus (Nervous system disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Fever (Infections and infestations) | 1 (2)
Hyponatremia (Nervous system disorders) | 1 (2)
Hypokalemia (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated due to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT04837131/Prot_SAP_000.pdf